CLINICAL TRIAL: NCT07264270
Title: A Phase 1, Randomized, Double-Blind, Single Dose Escalation Study to Assess the Safety and Tolerability of Transforaminal Epidural Administration of C-1101 Versus Sterile Saline in Adults With Chronic Painful Lumbosacral Radiculopathy
Brief Title: Study to Evaluate Safety of C-1101 Versus Sterile Saline in Adults With Chronic Painful Lumbosacral Radiculopathy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Consano Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: C-1101-101
Record Dates: First submitted 2025-11-20; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Lumbosacral Radicular Pain; Sciatic Radiculopathy; Sciatic Leg Pain; Sciatica; Lumbosacral Radicular Syndrome; Lumbosacral Radiculopathy
Keywords: Sciatica; Sciatic Nerve Pain; LSR; back pain; Lumbosacral Radiculopathy; Chronic Painful Lumbosacral Radiculopathy; non-opioid pain medication; transforaminal epidural injection
MeSH Terms: conditions — Sciatica; Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 - Low dose (Experimental)
  Interventions: Drug: C-1101; Other: Placebo: Sterile Saline
- Cohort 2 - Mid dose (Experimental)
  Interventions: Drug: C-1101; Other: Placebo: Sterile Saline
- Cohort 3 - High dose (Experimental)
  Interventions: Drug: C-1101; Other: Placebo: Sterile Saline

INTERVENTIONS:
Drug: C-1101 — C-1101
Other: Placebo: Sterile Saline — Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of C-1101 administered as a single dose, transforaminal epidural injection compared to sterile saline

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of painful LSR (sciatica) radiating to or below the knee, with an inadequate response to conservative care
* Body mass index < 35 kg/m2.

Exclusion Criteria:

* Presence of clinically significant disease or any other painful condition that may interfere with assessments.
* Any condition that currently requires blood or platelet transfusions.
* Diagnosed with schizophrenia, bipolar disorder, or major depressive disorder.
* Increased risk of bleeding or is taking anticoagulants or platelet aggregation inhibitors.
* History or presence of autonomic neuropathy, diabetic neuropathy, or other peripheral neuropathies.
* History of myocardial infarction within the last 6 months or congestive heart failure.
* The presence of an active malignancy or tumor.
* Have undergone a surgical procedure for back pain.
* Recent use of immunosuppressants, oral steroids, or intravenous steroids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events (TEAEs) | From Day 1 to Week 24
Incidence and severity of adverse events of special interest (AESIs) | From Day 1 to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Consano Chief Medical Officer, Study Director — Consano Bio
Locations (3):
- Australia (3):
  - Consano Bio Research Site, Broadmeadow, New South Wales
  - Consano Bio Research Site, Wahroonga, New South Wales
  - Consano Bio Research Site, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No